CLINICAL TRIAL: NCT07233694
Title: The Effects of Cold Spray and Stress Ball Methods on Perceived Pain, Comfort, and Satisfaction During Intramuscular Injection: A Randomized Controlled Trial
Brief Title: IM İnjection-PAIN-Cold Spray and Stress Ball
Acronym: CSB-PAIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, handan aydın kahraman, Asistant Professör, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Handan 1
Record Dates: First submitted 2025-06-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pain, Procedural; Acute Pain; Injection Site
Keywords: muscle intramuscular injection; Nursing; Nursing practice; Pain; stress ball; cold spray
MeSH Terms: conditions — Pain, Procedural; Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: The research was planned as a single-blind, randomized controlled experimental study.
Who Masked: Participant
Masking Description: The personnel responsible for drug administration are unaware of the treatment group allocations.
  Apart from the parties mentioned above, no further blinding was implemented
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No additional intervention will be applied to the participants in this group; only the standard IM injection protocol will be followed.
- Cold Spray Group (Experimental): Prior to the injection, cold spray was applied to an approximately 10 cm² area at the planned injection site from a distance of 15 cm for a duration of 5 seconds. Following this procedure, the intramuscular (IM) injection was administered within 15 seconds, and the entire process was completed in accordance with the standard protocol
  Interventions: Procedure: cold spray gruop
- Stress Ball Group (Experimental): Participants in this group were informed in advance about how to use the stress ball. After the ventrogluteal (VG) injection site was randomly selected, a medium-firm stress ball was placed in the hand on the non-injection side. Participants were instructed to rhythmically squeeze and release the ball throughout the procedure. The injection was then administered according to the predetermined standard protocol
  Interventions: Procedure: stress ball gruop

INTERVENTIONS:
Procedure: cold spray gruop — Arm Description: Before skin cleansing; cooling spray will be applied to a 10 cm2 area in the injection area from a distance of 15 cm for 5 seconds and diclofenac sodium injection will be applied within 15 seconds (Çetin and Avşar, 2022; Cevheroğlu and Büyükyılmaz, 2023). • IM injection protocol will be followed.
  Arms: Cold Spray Group
Procedure: stress ball gruop — The patients in the group will first be told how to use the ball. After the VG area to be injected is determined, a stress ball will be given to the patient's hand opposite the injection area and they will be asked to squeeze and loosen the ball. They will be told to repeat this until the procedure is completed.
  Arms: Stress Ball Group

SUMMARY:
Brief Summary:

Intramuscular (IM) injection is a widely used method for drug administration, with over 12 billion applications globally each year. Despite its therapeutic advantages, IM injection often causes pain, which can negatively impact patient comfort and lead to injection fear, non-compliance, and avoidance of healthcare services. Effective pain management during IM injection is an ethical and professional responsibility for nurses. This randomized controlled study aims to compare the effectiveness of cold spray and stress ball squeezing methods against standard practice in reducing IM injection-related pain. The study will be conducted in the emergency department of a university hospital in Turkey between March and June 2025, involving 66 patients prescribed IM diclofenac sodium. Participants will be randomly assigned to one of three groups: cold spray, stress ball, or control. Pain will be assessed using the Visual Analog Scale (VAS) within the first minute after injection.

DETAILED DESCRIPTION:
Study Description

Brief Summary:

Intramuscular (IM) injection is a widely used method for drug administration, with over 12 billion applications globally each year. Despite its therapeutic advantages, IM injection often causes pain, which can negatively impact patient comfort and lead to injection fear, non-compliance, and avoidance of healthcare services. Effective pain management during IM injection is an ethical and professional responsibility for nurses. This randomized controlled study aims to compare the effectiveness of cold spray and stress ball squeezing methods against standard practice in reducing IM injection-related pain. The study will be conducted in the emergency department of a university hospital in Turkey between March and June 2025, involving 66 patients prescribed IM diclofenac sodium. Participants will be randomly assigned to one of three groups: cold spray, stress ball, or control. Pain will be assessed using the Visual Analog Scale (VAS) within the first minute after injection.

Detailed Description:

Intramuscular (IM) injection is a fundamental method for delivering drugs directly into muscle tissue for systemic circulation. It is one of the most common invasive procedures in clinical practice globally, with over 12 billion applications annually. While offering faster absorption and higher bioavailability compared to oral and other parenteral routes for various pharmacological agents like vaccines, analgesics, sedatives, and antibiotics, IM injection can cause pain during administration, affecting patient comfort. This pain is a frequently reported side effect and can lead to injection phobia, non-adherence to treatment, and avoidance of health services. Consequently, managing pain during IM injections is a crucial ethical and professional responsibility for nurses.

Various non-pharmacological methods have been developed in nursing practice to reduce IM injection pain, and their efficacy has been extensively evaluated. These interventions include ShotBlocker, manual pressure, acupuncture, air-lock, distraction, and cold application. Cold application is a commonly preferred method for acute pain management due to its non-pharmacological effect and ease of clinical application. Cold sprays, in particular, offer significant advantages in clinical practice due to their minimal preparation, rapid effect, and low cost. These medical agents, derived from liquefied gases, rapidly evaporate from the skin surface, reducing local temperature and providing temporary superficial anesthesia. Their analgesic effects are achieved by inhibiting the activation of ion channels involved in pain transmission or by reducing the sensitivity of pain receptors. Limited studies have investigated cold spray use for IM injection pain control in adults. Comparative studies with ShotBlocker have reported that cold spray significantly reduces pain, but no significant difference was found between the two methods.

Distraction methods are effective nursing approaches that aim to reduce pain perception by shifting cognitive focus away from painful stimuli. The stress ball squeezing method, used within this strategy, has been applied in various invasive procedures and found effective in pain control. However, only one study has specifically evaluated its effect on IM injection pain. This study, conducted during Pfizer-BioNTech COVID-19 vaccination, reported no statistically significant effect of stress ball squeezing on pain levels.

Despite numerous studies on IM injection-related pain, it remains a prevalent clinical issue. Cold spray and stress ball squeezing offer practical options for pain reduction. However, studies evaluating their direct effects on IM injection pain are limited, and no direct comparative studies exist. Addressing this gap is crucial for evidence-based nursing care and improving patient experience.

This study aims to develop effective and applicable strategies to enhance care quality by comparatively evaluating cold spray, stress ball, and standard practice for reducing IM injection-related pain. Specifically, it aims to compare the effects of cold spray and stress ball squeezing methods on injection pain during IM injection and to examine their effectiveness in reducing pain compared to standard practice.

The research hypotheses are:

H1. The application of cold spray to the injection site during IM injection reduces the intensity of pain caused by the injection.

H2. Squeezing a stress ball during IM injection reduces the intensity of pain caused by the injection.

H3. Cold spray application is more effective than stress ball squeezing in reducing injection pain.

Study Design and Participants:

This study is a three-arm parallel-group, single-blind, randomized controlled experimental design, conducted in accordance with the CONSORT 2010 guidelines. The research will be conducted from March to June 2025 in the emergency department of a university hospital in Turkey. The sample will consist of 66 patients who present to the emergency department and have been prescribed IM diclofenac sodium. The sample size was calculated using G Power 3.1.9.7, based on variance values from a relevant article, with a 95% confidence interval, 0.05 error rate, 80% power, and an effect size of d=0.63, determining 22 participants per group.

Randomization and Allocation Concealment:

Participants will be randomly assigned to the cold spray, stress ball, or control group using a random number table generated via

https://www.random.org. Numbers from 1 to 66 will be written on separate slips of paper, placed in opaque envelopes, and sealed. Each eligible participant who consents to the study will select an envelope, and the number drawn will determine their group assignment.

Data Collection Instruments:

Data will be collected using a Patient Identification Form and a Visual Analog Scale (VAS). The Patient Identification Form will gather sociodemographic and clinical information such as age, gender, marital status, education level, body mass index, and chronic health conditions. The VAS is a valid and reliable 10-centimeter linear scale used to assess pain intensity, ranging from "no pain at all" (0) to "unbearable pain" (10). It is widely used in clinical studies due to its ease of application and effectiveness in evaluating pain reduction methods.

Intervention Materials:

Cold Spray: Galena® brand, aerosol form, containing butane, propane, and isobutane, which rapidly evaporates to reduce skin temperature and provide temporary superficial anesthesia.

Stress Ball: Approximately 10 cm in diameter, medium firmness, made of high-quality silicone, designed to change shape when squeezed and return to its original form.

Data Collection Process:

Before data collection, eligible patients will be informed about the study's purpose and content, and written and verbal consent will be obtained. All participants will complete the "Patient Identification Form" before the intervention. All IM injections will be administered by the same researcher following a standardized protocol to minimize variability. The injection side (right or left ventrogluteal region) will be randomly determined for each participant. Pain assessment will be performed within the first minute after injection by an independent nurse blinded to the patient's group, using the VAS.

Standard Intramuscular Injection Protocol:

Drug: Diclofenac sodium (3 mL)

Needle size: 21 Gauge

Syringe volume: 5 mL

Injection site: Left or right ventrogluteal region

Skin cleansing: The injection site will be cleaned with an alcohol swab in a 5 cm diameter, using circular movements from inside to outside, and 5 seconds will be waited for the area to dry before needle insertion.

Air-lock: 0.2-0.3 mL

Insertion angle: 90∘

Aspiration: Yes (5 sec)

Drug injection duration: 30 sec (1 mL / 10 sec)

Waiting time before needle removal: 10 sec

Post-injection application: Light pressure will be applied to the area for 15-20 seconds.

Pain measurement: Pain level will be assessed with VAS within the first 1 minute after injection and recorded.

Intervention Groups:

Cold Spray Group: Before the injection, cold spray will be applied for 5 seconds from a distance of 15 cm to an approximately 10cm 2 area at the planned injection site. The IM injection will then be performed within 15 seconds, following the standard protocol.

Stress Ball Group: Participants will be instructed on how to use the stress ball. After the injection site is randomly determined, a medium-firm stress ball will be given to the participant's non-injection hand, and they will be asked to rhythmically squeeze and release it throughout the procedure. The injection will be performed according to the standard protocol.

Control Group: Participants in this group will receive only the standard IM injection protocol without any additional interventions.

Ethical Considerations:

Ethical approval was obtained from Gümüşhane University Scientific Research and Publication Ethics Committee (2024, E-95674917-108.99-291198) and written application permission from Van Provincial Health Directorate before data collection. Informed written and verbal consent will be obtained from all participants after explaining the study's purpose and content. Principles of informed consent, respect for participant autonomy, and confidentiality of personal information will be maintained during data collection. All participants will be informed of their right to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years

Receiving intramuscular injection

Voluntarily agreed to participate in the study

Exclusion Criteria:

Skin disease at the injection site

Allergy to cold spray

Cognitive impairment preventing cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Intensity Using the Visual Analog Scale (VAS) Following a Cold Spray Intervention | Immediately after intramuscular injection (0-5 minutes)
  Pain intensity will be measured using the Visual Analog Scale (VAS). The VAS is a 100-millimeter horizontal line where 0 mm represents 'no pain' and 100 mm represents 'the worst imaginable pain'. A lower score on the VAS indicates a better outcome (less pain).
Assessment of Pain Intensity Using the Visual Analog Scale (VAS) During a Stress Ball Intervention | During intramuscular injection
  Squeezing a stress ball during intramuscular (IM) injection reduces the intensity of injection-related pain. Pain will be measured using the VAS.

SECONDARY OUTCOMES:
Comparison of Pain Intensity Scores Between the Cold Spray and Stress Ball Intervention Groups | Immediately after intramuscular injection (0-5 minutes)
  The mean pain scores, as measured by the Visual Analog Scale (VAS), will be compared between the group receiving the cold spray intervention and the group using the stress ball. The VAS is a 100-millimeter horizontal line where 0 mm represents 'no pain' and 100 mm represents 'the worst imaginable pain'. A lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Handan AYDIN KAHRAMAN, PHD, Principal Investigator — Erzincan Binali Yildirim Universitesi
Locations (1):
- Erzincan Binali Yıldırım University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional data protection policies. The data collected in this study are intended solely for the purposes of this specific research.

REFERENCES:
- [Result] Ayinde O, Hayward RS, Ross JDC. The effect of intramuscular injection technique on injection associated pain; a systematic review and meta-analysis. PLoS One. 2021 May 3;16(5):e0250883. doi: 10.1371/journal.pone.0250883. eCollection 2021. PMID 33939726
- [Result] Basak T, Demirtas A, Yorubulut SM. Virtual reality and distraction cards to reduce pain during intramuscular benzathine penicillin injection procedure in adults: A randomized controlled trial. J Adv Nurs. 2021 May;77(5):2511-2518. doi: 10.1111/jan.14782. Epub 2021 Feb 19. PMID 33608955
- [Result] Cmc S, Lord H, Vargese SS, Kurian N, Cherian SA, Mathew E, Fernandez R. Effectiveness of physical stimulation for reducing injection pain in adults receiving intramuscular injections: a systematic review and meta-analysis. JBI Evid Synth. 2023 Feb 1;21(2):373-400. doi: 10.11124/JBIES-20-00590. PMID 36758552

DOCUMENTS (3):
  • Study Protocol (2025-10-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT07233694/Prot_000.pdf
  • Statistical Analysis Plan: Statistical (2025-10-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT07233694/SAP_001.pdf
  • Informed Consent Form (2025-10-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT07233694/ICF_002.pdf